CLINICAL TRIAL: NCT07302945
Title: High-Resolution Immune Dynamics Following OTS-412 Oncolytic Vaccinia Virus Administration in a Healthy Volunteer(Self-experiment)
Brief Title: A Single-volunteer Study of Immune Response Following OTS-412 Vaccinia Virus Systemic Injection(Self-experiment)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bionoxx Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OTS412-HV
Record Dates: First submitted 2025-11-16; First posted 2025-12-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OV Treated healthy arm (Experimental)
  Interventions: Biological: OTS-412

INTERVENTIONS:
Biological: OTS-412 — After hospitalization, OTS-412 was infused for one hour.

SUMMARY:
Following oncolytic virus (OV) administration, the host immune response is initiated immediately and evolves dynamically. However, in clinical OV therapy, it is virtually impossible to capture these immune events in real time. To address this gap, the principal investigator conducted a high-resolution immune monitoring study in a healthy volunteer.

ELIGIBILITY:
Inclusion Criteria:

* A healthy adult

Exclusion Criteria:

* N/A

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Changes in ANC(absolute neutrophil count) over time | 4 hour, 8 hour, 20 hour, 24 hour, Day 2, Day 5, Day 8, Day 16
Changes in lymphocytes count over time | 4 hour, 8 hour, 20 hour, 24 hour, Day 2, Day 5, Day 8, Day 16

SECONDARY OUTCOMES:
FLow cytometry | 4 hour, 8 hour, 20 hour, 24 hour, Day 2, Day 5, Day 8, Day 16
  CD surface subtyping for each sampling

OTHER OUTCOMES:
Measurement of GFP expressing neutrophils following ex vivo infection with gfp report viral vector combined with CD surface phenotypes. | 4 hour, 48 hour, Day 8, Day 16

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Medical college, Busan, South Korea